CLINICAL TRIAL: NCT06428916
Title: The Effect of Facilitated Tucking Position During Endotracheal Suctioning on Physiological Measurement and Behavioral Responses of the Preterm Neonates
Brief Title: Facilitated Tucking Position During Endotracheal Suctioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Wardany Abdelaal Mohamed, assistant professor of pediatric nursing, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KafrelsheikhU2
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: Physiological measurement; Behavioral Responses of the Preterm Neonates; Facilitated Tucking Position; Endotracheal Suctioning
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Consisted of 20 neonates who will receive tucking position during endotracheal suctioning
  Interventions: Procedure: tucking position during endotracheal suctioning
- Control group (No Intervention): Consisted of 20 neonates who will receive routine care during Endotracheal suctioning

INTERVENTIONS:
Procedure: tucking position during endotracheal suctioning — , the staff nurse will perform the endotracheal suctioning while the researcher will carried out the intervention
  Arms: Study Group

SUMMARY:
Aim of the present study The present study will aimed to determine the effect of facilitated tucking position during endotracheal suctioning on physiological criteria and behavioural responses of the preterm neonates.

Research Hypotheses

1. Preterm neonates who receive facilitated tucking position during endotracheal suctioning exhibit more stable physiological criteria than those who do not.
2. Preterm neonates who receive facilitated tucking position during endotracheal suctioning exhibit more stable behavioral responses than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 32 and 36 weeks, weight 1200 grams or greater.
* Postnatal age: two days after delivery to allow for resolution of analgesia or anesthesia received by their mothers during labor.
* Have endotracheal intubation.

Exclusion Criteria:

* Preterm neonates who have congenital anomalies or neurological malformations, intracranial hemorrhage, seizures.
* Preterm neonates who received sedatives within four hours before the intervention
* Preterm neonates who exposed to any uncomfortable procedure for at least 30 minutes prior to the intervention.

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of heart rate of preterm neonates on Neonates' Physiological Assessment Tool during and immediately following the endotracheal suction procedure | during procedural and immediately after procedure
  Neonates' Physiological Assessment Tool was developed by researchers after a review of relevant literature to assess Physiological Parameters of preterm neonates as Heart Rate (HR)
Change from baseline of Respiratory Rate of preterm neonates on Neonates' Physiological Assessment Tool during and immediately following the endotracheal suction procedure | during procedural and immediately after procedure
  Neonates' Physiological Assessment Tool was developed by researchers after a review of relevant literature to assess Physiological Parameters of preterm neonates as Respiratory Rate (RR)
Change from baseline of oxygen saturation in blood of preterm neonates on Neonates' Physiological Assessment Tool during and immediately following the endotracheal suction procedure | during procedural and immediately after procedure
  Neonates' Physiological Assessment Tool was developed by researchers after a review of relevant literature to assess Physiological Parameters of preterm neonates as oxygen saturation in blood(SPO2)

SECONDARY OUTCOMES:
change of baseline of Neonates' behavioral states on Anderson Behavioral State Scale during and immediately following the endotracheal suction procedure | during procedural and immediately after procedure
  This scale was adopted from Anderson et al.(1990) to assess the behavioral organization of preterm neonates. Neonates' behavioral states are assessed by observing their respiratory regularity, opening or closing of the eyes, limb and trunk activity, and the intensity of crying. Based on the observations, the scale will differentiate 12 behavioral states, including; regular quiet sleep (1), irregular quiet sleep (2), active sleep (3), very active sleep (4), drowsy (5), alert inactivity (6), quite awake (7), active awake (8), very active awake (9), fussing (10), crying (11) and hard crying (12). Scores from 1 to 5 indicate that the neonate is sleeping. Scores from 6 to 8 indicate that the neonate is awake and calm. Scores from 9 to 12 indicate that the neonate is in a state of restless activity or fussiness, which takes substantial energy

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No